CLINICAL TRIAL: NCT00760370
Title: Bone Retention of Bisphosphonate (Zometa) in Patients With Multiple Myeloma or Breast Cancer With Metastases to Bone
Brief Title: Comparison of Zometa Retention and Effect in Multiple Myeloma and Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Odense University Hospital (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-003777-13; 2007-003777-13
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Multiple Myeloma; Breast Cancer
Keywords: bone marker; bisphosphonate; Zometa; retention; breast cancer; multiple myeloma; CTX; bone specific ALP
MeSH Terms: conditions — Multiple Myeloma; Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Zoledronic Acid — 4 mg intravenous (iv), one treatment
  Other Names: Zometa

SUMMARY:
The investigators major aim is to determine whether there is a difference in the retention of zoledronic acid in multiple myeloma patients, compared to patients with breast cancer metastasis to bone. In addition the investigators wish to analyze if the retention of zoledronic acid is correlated to the extent of bone resorption/formation, and if there is a tendency to changes in retention with sequential treatment.

DETAILED DESCRIPTION:
The clinical benefit from treatment with bisphosphonates has been documented in a large number of clinical studies, and bisphosphonates are now widely used for treatment of pain and prevention of bone fractures or vertebral collapse for example in patients with cancer metastasis to bone or multiple myeloma.

Repeated intravenous administration of the more potent bisphosphonates (pamidronate and zoledronic acid) are often used for treatment of osteolytic disease caused by disseminated cancer or multiple myeloma, while the less potent oral bisphosphonates are often prescribed for treatment of benign osteoporosis. The recommended dose and time schedule for treatment with the more potent bisphosphonates is based on concerns of avoiding toxicity and at the same time obtaining maximal clinical benefit. Clinical studies in multiple myeloma and bone metastasis show significant activity of pamidronate (90 mg by iv infusion during 2-4 hours) or zoledronic acid (4 mg iv during 15 min) repeated every 4 weeks after a treatment period of 9 months and beyond, but the optimal duration of treatment is not known. This is a particular important issue since the use of potent bisphosphonates have been brought in connection with osteonecrosis.

In the present study we will compare the retention of Zometa with the effect on bone markers in patients with multiple myeloma or breast cancer with metastases to bone.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer and metastases to bone.
* Patients diagnosed with multiple myeloma.
* Patients who are scheduled to receive Zometa.
* Post-menopausal women (at least 10 months since last period).
* Newly diagnosed patients must have clear signs of osteolysis.

Exclusion Criteria:

* Anti-estrogen treatment.
* Patients given chemotherapy during or less than 7 days before study begin.
* Patients receiving glucocorticoids less than 5 days prior to study begin or during the study period (14 days)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Amount of Zometa retained in body | 48 hrs

SECONDARY OUTCOMES:
Changes in bone markers | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Torben Plesner, MD, PhD, Principal Investigator — Vejle Hospital
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle

REFERENCES:
- [Background] Cremers SC, Papapoulos SE, Gelderblom H, Seynaeve C, den Hartigh J, Vermeij P, van der Rijt CC, van Zuylen L. Skeletal retention of bisphosphonate (pamidronate) and its relation to the rate of bone resorption in patients with breast cancer and bone metastases. J Bone Miner Res. 2005 Sep;20(9):1543-7. doi: 10.1359/JBMR.050522. Epub 2005 May 31. PMID 16059626